CLINICAL TRIAL: NCT05061082
Title: Genomic Evolution of Metastasis in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 80/GCN-HDDD 2021
Record Dates: First submitted 2021-09-09; First posted 2021-09-29 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Gastric Cancer; Metastasis
Keywords: Gastric Cancer; Metastasis
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to track tumor evolution of regional and distant metastases in gastric cancer using the Next Generation Sequencing technologies.

DETAILED DESCRIPTION:
Gastric cancer is the fourth most common cancer in Vietnam with high mortality rate. Metastasis is the leading cause of death in gastric cancer patients, with median overall survival of less than 1 year. Currently, there is no effective treatment because the molecular mechanism of metastasis remains unclear. The aim of this study is to use advanced NGS technologies to dissect the genomic changes (genetic, epigenetic and transcriptional changes) of the primary tumor and associated metastatic sites of the same patients. With that, the investigators can reconstruct the clonal evolution from primary tumor to metastasis, identify key pathways governing metastasis development that can be targeted for future therapeutic development.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged 18 years and older
2. Histologically proven primary gastric adenocarcinoma and clinical evidence of metastasis (N1-3M1)
3. Biopsies can be taken at multiple sites
4. No known other concomitant cancer diagnosis
5. Signed informed consent

Exclusion Criteria:

1. Gastric adnocarcinoma cannot be confirmed primary
2. Unable to undergo biopsy or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic gastric adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Genetic and epigenetic changes of the tumor | 3 months after surgery
  Ultra-deep NGS of the primary tumor and associated metastatic sites from the same patients to identify mechanism governing metastasis development

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No